CLINICAL TRIAL: NCT03437083
Title: A Nationwide, Multi-institutional Retrospective Study of Efficacy and Safety of Eribulin in Korean Breast Cancer Patients
Brief Title: A Study to Investigate the Efficacy and Safety of Eribulin in Korean Breast Cancer Participants
Status: Completed | Type: Observational
Sponsor: Eisai Korea Inc. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: E7389-M082-602
Record Dates: First submitted 2018-01-08; First posted 2018-02-19 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2018-06

CONDITIONS: Locally Advanced or Metastatic Breast Cancer
Keywords: Breast neoplasms; Metastatic breast cancer; E7389
MeSH Terms: conditions — Breast Neoplasms | interventions — eribulin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Eribulin: Eribulin was administered at a dose of 1.4 milligrams per meters squared (mg/m^2) (as eribulin 1.23 mg/m^2) by a 2- to 5-minute intravenous infusion or as a diluted solution on Day 1 and Day 8 every 21 days.
  Interventions: Drug: Eribulin mesylate

INTERVENTIONS:
Drug: Eribulin mesylate — intravenous infusion
  Other Names: Halaven; E7389

SUMMARY:
The primary objective of the study is to observe efficacy in terms of progression-free survival rate at 6 months in eribulin-treated breast cancer participants retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of locally advanced or metastatic breast cancer
* Participants who were treated with Eribulin between 01 June, 2014 and 31 December, 2016

Exclusion Criteria:

* Not applicable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male and female participants diagnosed with locally advanced or metastatic breast cancer, who had experience with eribuin-treatment
Sampling Method: Probability Sample
Enrollment: 340 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) rate at 6 months | 6 months
  PFS rate at 6 months is estimated based on the tumor response evaluation and is defined as the proportion of participants alive and progression-free at 6 months from the initial treatment of eribulin.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | From the start date of therapy with eribulin to the date of disease progression or death from any cause (1 day to up to approximately 2 years)
  PFS is defined as the time from the start date of therapy with eribulin to the date of disease progression or death from any cause. Participants without progression will be censored, progression free at the date of late follow-up.
Overall Survival (OS) | From the start date of therapy with eribulin to the date of death from any cause or last follow-up (1 day to up to approximately 2 years)
  OS is defined as the time from the start date of therapy with eribulin to the date of death from any cause or last follow-up.
Time to treatment failure (TTF) | From the first treatment with eribulin to discontinuation of treatment for any reason (1 day to up to approximately 2 years)
  TTF is defined as a time from first treatment with eribulin to discontinuation of treatment for any reason, including disease progression, treatment toxicity, and death.
Tumor response rate (TRR) | From the start date of therapy with eribulin to the date of death from any cause or last follow-up (1 day to up to approximately 2 years)
  TRR will be evaluated by medical records. ORR is defined as the sum of obtained PR and CR and the clinical benefit rate (CBR) is defined as the sum of PR, CR and stable disease (SD) maintained for at least six months. Disease control rate (DCR) is defined as the sum of PR, CR and SD.
Number of participants with any treatment-emergent adverse event (TEAE) | 6 months
  An adverse event (AE) is any untoward medical occurrence in a participant or clinical investigation participant administered an investigational product. An AE does not necessarily have a causal relationship with the medicinal product. A TEAE is defined as an AE that emerges during treatment, having been absent at pretreatment (baseline) or (1) reemerges during treatment, having been present at pretreatment (baseline) but stopped before treatment, or (2) worsens in severity during treatment relative to the pretreatment state, when the AE is continuous.
PFS in eribulin-treated breast cancer participants according to line of treatment for advanced disease and tumor subtype (receptor status and molecular subtype) | From the start date of therapy with eribulin to the date of disease progression or death from any cause (1 day to up to approximately 2 years)
  PFS is defined as the time from the start date of therapy with eribulin to the date of disease progression or death from any cause. Participants without progression will be censored, progression free at the date of late follow-up.
OS in eribulin-treated breast cancer participants according to line of treatment for advanced disease and tumor subtype (receptor status and molecular subtype) | From the start date of therapy with eribulin to the date of death from any cause or last follow-up (1 day to up to approximately 2 years)
  OS is defined as the time from the start date of therapy with eribulin to the date of death from any cause or last follow-up.
TTF in eribulin-treated breast cancer participants according to line of treatment for advanced disease and tumor subtype (receptor status and molecular subtype) | From the first treatment with eribulin to discontinuation of treatment for any reason (1 day to up to approximately 2 years)
  TTF is defined as a time from first treatment with eribulin to discontinuation of treatment for any reason, including disease progression, treatment toxicity, and death.
TRR in eribulin-treated breast cancer participants according to line of treatment for advanced disease and tumor subtype (receptor status and molecular subtype) | From the start date of therapy with eribulin to the date of death from any cause or last follow-up (1 day to up to approximately 2 years)
  TRR will be evaluated by medical records. ORR is defined as the sum of obtained PR and CR and the CBR is defined as the sum of PR, CR and SD maintained for at least six months. DCR is defined as the sum of PR, CR and SD.
PFS rate in eribulin-treated breast cancer participants comparing early (≤ third line) to late (≥ fourth line) use | From the start date of therapy with eribulin to the date of disease progression or death from any cause (1 day to up to approximately 2 years)
  PFS is defined as the time from the start date of therapy with eribulin to the date of disease progression or death from any cause. Participants without progression will be censored, progression free at the date of late follow-up.
OS in eribulin-treated breast cancer participants comparing early (≤ third line) to late (≥ fourth line) use | From the start date of therapy with eribulin to the date of death from any cause or last follow-up (1 day to up to approximately 2 years)
  OS is defined as the time from the start date of therapy with eribulin to the date of death from any cause or last follow-up.
TTF in eribulin-treated breast cancer participants comparing early (≤ third line) to late (≥ fourth line) use | From the first treatment with eribulin to discontinuation of treatment for any reason (1 day to up to approximately 2 years)
  TTF is defined as a time from first treatment with eribulin to discontinuation of treatment for any reason, including disease progression, treatment toxicity, and death.
TRR in eribulin-treated breast cancer participants comparing early (≤third line) to late (≥ fourth line) use | From the start date of therapy with eribulin to the date of death from any cause or last follow-up (1 day to up to approximately 2 years)
  TRR will be evaluated by medical records. ORR is defined as the sum of obtained (PR) and CR and the CBR is defined as the sum of PR, CR and SD maintained for at least 6 months. DCR is defined as the sum of PR, CR and SD.
Number of participants with the indicated action to TEAEs | 6 months
  An AE is any untoward medical occurrence in a participant or clinical investigation participant administered an investigational product. An AE does not necessarily have a causal relationship with the medicinal product. A TEAE is defined as an AE that emerges during treatment, having been absent at pretreatment (baseline) or (1) reemerges during treatment, having been present at pretreatment (baseline) but stopped before treatment, or (2) worsens in severity during treatment relative to the pretreatment state, when the AE is continuous.
Number of participants with TEAEs resulting in discontinuation of eribulin | 6 months
  An AE is any untoward medical occurrence in a participant or clinical investigation participant administered an investigational product. An AE does not necessarily have a causal relationship with the medicinal product. A TEAE is defined as an AE that emerges during treatment, having been absent at pretreatment (baseline) or (1) reemerges during treatment, having been present at pretreatment (baseline) but stopped before treatment, or (2) worsens in severity during treatment relative to the pretreatment state, when the AE is continuous.
Number of participants using supportive drugs to treat AEs | 6 months
  Treatment of adverse events will be collected retrospectively.
Median number of eribulin cycles | 6 months
  Data will be collected to observe a treatment pattern of eribulin in the real world.
Number of participants experiencing a dose reduction | 6 months
  Data will be collected to observe a treatment pattern of eribulin in the real world.
Mean duration of treatment | 6 months
  Duration of treatment is defined as the time from documentation of the start of eribulin treatment to the date of permanent discontinuation.
Mean duration of response | 6 months
  Duration of response is defined as the time from the first documented evidence of CR or PR (whichever status is recorded first) until the first documented sign of disease progression or death due to any cause.
Mean dose intensity | 6 months
  Dose intensity is defined as the amount of drug milligrams per meters squared (mg/m^2) delivered to a participant in a week of treatment.
Number of participants with the indicated reason for treatment discontinuation | 6 months
  Data will be collected to observe a treatment pattern of eribulin in the real world.

CONTACTS AND LOCATIONS:
Locations (14):
- South Korea (14):
  - Eisai Trial site_03, Ansan
  - Eisai Trial site_04, Busan
  - Eisai Trial site_05, Busan
  - Eisai Trial site_06, Busan
  - Eisai Trial site_09, Daegu
  - Eisai Trial site_13, Daejeon
  - Eisai Trial site_14, Gwangju
  - Eisai Trial site_01, Seoul
  - Eisai Trial site_02, Seoul
  - Eisai Trial site_07, Seoul
  - Eisai Trial site_10, Seoul
  - Eisai Trial site_11, Seoul
  - Eisai Trial site_12, Seoul
  - Eisai Trial site_08, Suwon